CLINICAL TRIAL: NCT04370639
Title: Non-Invasive Hemorrhage Monitoring: A Pilot Study to Assess the Feasibility and Tolerability of the AccuFlow Perfusion Sensor for the Detection of Intrapartum Hemorrhage
Brief Title: A Pilot Study to Assess the Feasibility and Tolerability of the AccuFlow Perfusion Sensor for Intrapartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Megan Lord (Other)
Collaborators: ThermaSENSE Corp (Unknown)
Responsible Party: Sponsor-Investigator, Megan Lord, Principal Investigator, Women and Infants Hospital of Rhode Island
Organization: Women and Infants Hospital of Rhode Island (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1498912
Record Dates: First submitted 2020-04-27; First posted 2020-05-01 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Hemorrhage, Postpartum; Hemorrhage; Vasoconstriction
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- AccuFlow Sensor (Experimental): These 50 patients will wear the AccuFlow sensor device during their surgery, and will complete the post-procedural survey. The data will be reviewed after 25 patients, and the pilot study may be stopped at that point if it is felt that the device feasibility and tolerability have been adequately established.
  Interventions: Device: AccuFlow sensor; Other: Survey

INTERVENTIONS:
Device: AccuFlow sensor — AccuFlow sensor will be worn and survey completed
Other: Survey — Patients will be asked to complete a survey regarding device tolerability after completing their cesarean section.

SUMMARY:
Obstetric hemorrhage is one of the leading causes of maternal death worldwide. One of the challenges in management of hemorrhage is that young, healthy women compensate for blood loss via peripheral vasoconstriction, so they maintain their blood pressure and heart rate at normal levels even after experiencing significant blood loss. By the time vital sign abnormalities appear, interventions must be performed extremely rapidly to avoid organ damage and maternal death. Clinical methods of estimating blood loss in real time, such as visual estimation, are notoriously unreliable, and changes in laboratory testing such as hemoglobin levels lag hours behind actual blood loss. A tool which can detect and quantify blood loss in real time, before vital sign changes occur, has the potential to allow for earlier mobilization of resources and intervention in these cases, thus saving lives. This device is meant to detect changes in skin blood flow which reflect vasoconstriction. The investigators believe that this device, therefore, has the potential to be able to detect and quantify blood loss in real-time. However, as this novel device has never been used for this purpose, before undertaking a large clinical trial, the investigators feel it is necessary to perform a pilot study to assess the feasibility and tolerability of this device. The investigators plan to test this by asking 50 patients undergoing planned cesarean section to wear the device during their surgery. The device will collect skin perfusion measurements during the surgery, which will not be available to the operating team. The patients will also be asked to complete a survey regarding their experience wearing the device. The investigators will use this information to ensure that the device is transmitting interpretable data, that patients feel the device is tolerable during surgery, and to ensure that the device can be used in the operating room without any unforeseen logistical challenges which would need to be addressed in planning a larger trial. The investigators will perform a preliminary comparison of sensor readings to laboratory findings, to assist in planning a larger trial.

DETAILED DESCRIPTION:
Hemorrhage remains the leading cause of direct pregnancy-related death in both the developing world and the developed world. Young, healthy patients compensate for hemorrhage via peripheral vasoconstriction, delaying the emergence of vital sign abnormalities until 15-30% of total blood volume has been lost (1-2L in a term pregnant patient). A significant drop in blood pressure and marked tachycardia (>120bpm) are not seen until 30-40% of blood volume has been lost. After 40% loss, however, patients may rapidly decompensate, leaving a narrow window between the emergence of vital sign abnormalities and rapid clinical decompensation. In facilities where obstetricians and anesthesiologists are not in-house at all times and blood product availability is limited, this narrow window may prove catastrophic.

Furthermore, management of obstetrical blood loss presents many unique challenges. First, during delivery, when hemorrhage is expected and occurs acutely and visibly, blood is often mixed with amniotic fluid, making it difficult to establish actual blood loss. Second, laboratory measurement of hemoglobin concentrations can be falsely normal during an acute episode of bleeding, as the hemoglobin measured does not reflect actual hemoglobin concentration until several hours after the hemorrhage event, when equilibration occurs. Third, unlike other surgical patients, postpartum women are expected to experience ongoing vaginal bleeding after their delivery. Bleeding which is persistently slightly heavier than average can lead to significant blood loss over a period of several days, without either the patient or the staff caring for her recognizing the hemorrhage until the patient becomes symptomatic or vital sign instability occurs. The postpartum uterus can serve as a reservoir for retained blood and clot, allowing a patient to continue bleeding into her uterus after delivery without any external evidence of bleeding. In a thin patient this is frequently recognized on "fundal checks" where the size of the uterus is evaluated, but in obese patients the uterine fundus may be difficult to appreciate, and a significant volume of blood can accumulate in the uterus before it is recognized.

Due to the high risk of mortality related to postpartum hemorrhage and the difficulties providers face quantifying blood loss accurately after delivery,, it is imperative to develop a tool that can detect and quantify hemorrhage before vital sign changes occur. This tool should be simple to use, allowing healthcare providers at all levels to identify hemorrhage early and to mobilize appropriate resources. This will facilitate earlier intervention to treat blood loss before clinical decompensation. As stated, vasoconstriction is the earliest physiologic responses to acute hypovolemia6 and, as such, would be an appropriate target for such a tool.

The AccuFlow Sensor is a device that is based on Combined Heat-Flux and Temperature Sensor (CHFT+) technology developed in the heat transfer laboratory at Virginia Tech and produced by ThermanSENSE Corp (Roanoke, VA). The device, which consists of a heat flux sensor, a thin-film thermocouple, and a heater element, makes direct, quantitative measurements of perfusion occurring at the surface of exposed tissue in real-time. The sensor is less than 1mm thick, covers one square inch of skin, and adheres to the patient's skin using a piece of medical-grade silicone adhesive tape. The heater applies a small amount of heat to the skin surface, raising its temperature to approximately 39 degrees C. The heat flux sensor measures the rate at which the heat dissipates into the tissue, and uses this to calculate perfusion using the Pennes Bio-Heat Transfer Equation, which was developed to describe patterns of heat distribution in the human forearm and which has been the standard tool to predict temperature distributions in living human tissue since the 1950s.10 The sensor measures both surface perfusion and deep perfusion (1-2cm below the skin surface).

The primary theoretical source of patient injury or discomfort from the device is thermal injury from the heater element. Under typical circumstances, the device heats up to approximately 39 degrees Celsius (102 Fahrenheit, the temperature of a typical hot tub), and to prevent thermal injury, the device automatically shuts off should it reach a temperature of 45 C (113F, just above the typical hot-shower temperature of 110F). The device has been tested for comfort and tolerability on 20 healthy volunteers, who reported no discomfort while wearing the device or afterwards. Prior studies have shown no evidence of thermal injury in tissues exposed to a temperature of 39C for prolonged periods, and that exposure to temperatures of 45C causes mild thermal injury only after 150 minutes of constant exposure.11 As this device only heats up while it is taking a measurement, and never higher than 45C, the risk of a thermal injury while wearing the device for the duration of a cesarean section as planned during this study is extremely low. However, should the sensor become uncomfortable to the patient, it can easily be removed. To date, the sensor has been used to evaluate viability of organs intended for transplantation, by measuring blood flow at the surface of the organ.7 Currently, the sensor is being used to evaluate differences in tissue perfusion between pediatric patients with sickle cell anemia and healthy controls in an ongoing research study at Virginia Tech. Of note, the device meets FDA criteria for a nonsignificant risk device, and has been determined to be a nonsignificant risk device by the Institutional Review Board at Virginia Tech/Carilion Clinic for use in adult and pediatric patients at Carilion Clinic facilities. As mentioned before, the patent-pending AccuFlow device is provided by ThermaSENSE Corp. (Roanoke, VA) and a number of sensors will be contributed for the purpose of this study. The device has not yet been studied for detection of obstetric hemorrhage.

In order to determine whether the device is able to accurately detect obstetric hemorrhage, it must be tested on a number of patients who can be identified and enrolled in a research study prior to experiencing a significant volume of blood loss, and whose volume of blood loss can be retrospectively calculated with some degree of accuracy and compared to the device's measurements. Patients undergoing planned, scheduled cesarean delivery are an ideal study population, because they undergo routine measurements of height, weight, hemoglobin, and hematocrit before surgery, and a repeat hemoglobin and hematocrit the day after surgery, once physiologic equilibration has occurred. From these hematocrit measurements, the percentage and volume of blood loss can be calculated and compared to the measurements obtained from the Non-Invasive Blood Perfusion Sensor.

The investigators propose to perform a pilot study consisting of 50 patients, with a planned interim analysis after 25 patients. These patients will be asked to wear the sensor during their planned cesarean delivery, and to complete a survey immediately after their surgery regarding their experience wearing the device. The device will be applied preoperatively and removed postoperatively, and a member of the study team will remain in the operating room to monitor the device and to note any significant events which occur during surgery, as well as any potential challenges with the use of the device which must be considered in planning future trials. Additional information will be gathered from the patients' charts including demographics, height, weight, hemoglobin and hematocrit before and after surgery. The investigators will review the sensor readings and the laboratory findings to determine which of a number of different methods of analyzing device readings should be used in a larger trial, as well as which of the measurement sites used by the sensors provides the most relevant data, in order to streamline the device design prior to a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* English speaking
* Undergoing planned cesarean section at Women and Infants Hospital
* BMI on admission less than or equal to 35 kg/m2
* Preoperative hemoglobin greater than or equal to 11.5g/dL on routine labs

Exclusion Criteria:

* History of allergy or other adverse reaction to adhesives
* Fever at the time of recruitment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Improving sensor design and analysis | 6 months
  We will use the sensor readings obtained from this study to determine how best to obtain and analyze sensor readings in a larger trial. This will include comparing different ratios of readings (both different points in time during the case and different measurement sites on the patient) to determine the ideal number and locations of sensors, and ideal method of data analysis, for a larger trial.

SECONDARY OUTCOMES:
Device Tolerability | 6 months.
  Patients will be asked to complete a survey after their cesarean rating the tolerability of the device, as well as the tolerability of standard anesthesia monitoring equipment (blood pressure cuff and pulse oximeter), to assess how the tolerability of the novel device compares to equipment already in use. This will be done in this way because although there is a validated scale for tolerability of wearable computer devices, this scale is only validated as a comparison between two options, and no absolute threshold below which a device is considered "tolerable" has been established.
Accuracy | 6 months
  We will compare the available device readings to the available lab measurements of hemorrhage, to determine if a difference is seen between patients with 10% blood volume lost vs 20% blood volume lost. This will assist in planning a larger trial by determining how many patients with higher-volume blood loss would need to be included, and therefore what total enrollment would likely be needed in the larger trial.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Lord, MD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women and Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, we do not plan to make IPD available.

REFERENCES:
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] LOW JA, JOHNSTON EE, MCBRIDE RL. BLOOD VOLUME ADJUSTMENTS IN THE NORMAL OBSTETRIC PATIENT WITH PARTICULAR REFERENCE TO THE THIRD TRIMESTER OF PREGNANCY. Am J Obstet Gynecol. 1965 Feb 1;91:356-63. doi: 10.1016/0002-9378(65)90250-4. No abstract available. PMID 14258262
- [Background] Mutschler M, Paffrath T, Wolfl C, Probst C, Nienaber U, Schipper IB, Bouillon B, Maegele M. The ATLS((R)) classification of hypovolaemic shock: a well established teaching tool on the edge? Injury. 2014 Oct;45 Suppl 3:S35-8. doi: 10.1016/j.injury.2014.08.015. PMID 25284231
- [Background] Chandra S, Tripathi AK, Mishra S, Amzarul M, Vaish AK. Physiological changes in hematological parameters during pregnancy. Indian J Hematol Blood Transfus. 2012 Sep;28(3):144-6. doi: 10.1007/s12288-012-0175-6. Epub 2012 Jul 15. PMID 23997449
- [Background] Ashok Y, Roy PS, Goyal BK. ACUTE NORMOVOLEMIC HEMODILUTION IN PATIENTS UNDERGOING ELECTIVE MAJOR SURGERY. Med J Armed Forces India. 2000 Jul;56(3):216-218. doi: 10.1016/S0377-1237(17)30170-3. Epub 2017 Jun 10. PMID 28790711
- [Background] Schiller AM, Howard JT, Convertino VA. The physiology of blood loss and shock: New insights from a human laboratory model of hemorrhage. Exp Biol Med (Maywood). 2017 Apr;242(8):874-883. doi: 10.1177/1535370217694099. Epub 2017 Jan 1. PMID 28346013
- [Background] O'Brien TJ, Roghanizad AR, Jones PA, Aardema CH, Robertson JL, Diller TE. The Development of a Thin-Filmed Noninvasive Tissue Perfusion Sensor to Quantify Capillary Pressure Occlusion of Explanted Organs. IEEE Trans Biomed Eng. 2017 Jul;64(7):1631-1637. doi: 10.1109/TBME.2016.2615241. Epub 2016 Oct 5. PMID 28113229
- [Background] Conner SN, Tuuli MG, Colvin R, Shanks AL, Macones GA, Cahill AG. Accuracy of Estimated Blood Loss in Predicting Need for Transfusion after Delivery. Am J Perinatol. 2015 Nov;32(13):1225-30. doi: 10.1055/s-0035-1552940. Epub 2015 May 22. PMID 26007310
- [Background] Sylla RR, Lee KL. Correlating Quantitative Blood Loss and Estimated Blood Loss With Postoperative Change in Hematocrit After Cesarean Delivery [258]. Obstetrics & Gynecology. 2015;125:83S. doi:10.1097/01.aog.0000463235.89427.b3
- [Background] PENNES HH. Analysis of tissue and arterial blood temperatures in the resting human forearm. J Appl Physiol. 1948 Aug;1(2):93-122. doi: 10.1152/jappl.1948.1.2.93. No abstract available. PMID 18887578
- [Background] Moritz AR, Henriques FC. Studies of Thermal Injury: II. The Relative Importance of Time and Surface Temperature in the Causation of Cutaneous Burns. Am J Pathol. 1947 Sep;23(5):695-720. No abstract available. PMID 19970955
- [Background] Knight JF, Baber C, Schwirtz A, Bristow HW. The comfort assessment of wearable computers. Proceedings Sixth International Symposium on Wearable Computers. doi:10.1109/iswc.2002.1167220